CLINICAL TRIAL: NCT03808870
Title: A Phase 1, Open-label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Efficacy of NBM-BMX in Asian Subjects With Advanced Solid Tumors
Brief Title: A Safety and Pharmacokinetic Study of NBM-BMX Administered Orally to Asian Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NatureWise Biotech & Medicals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBM-BMX-002
Record Dates: First submitted 2019-01-10; First posted 2019-01-18 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBM-BMX (Experimental)
  Interventions: Drug: NBM-BMX softgel capsules

INTERVENTIONS:
Drug: NBM-BMX softgel capsules — Patients will initially receive NBM-BMX orally once a day at 100 mg per day.

SUMMARY:
NBM-BMX is an orally available new chemical entity to inhibit HDAC8 activity specifically, being developed as a potential anti-cancer therapeutic by NatureWise. The objectives of this study are to evaluate the safety, pharmacokinetics, and preliminary efficacy of NBM-BMX as monotherapy in subjects with advanced solid tumors (Arm A) or in combination with the standard of care treatment (i.e., concomitant RT/TMZ followed by adjuvant TMZ) in subjects with newly diagnosed glioblastoma (Arm B).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced, non-resectable, and/or metastatic solid tumor refractory to standard of care therapy, or for whom no standard of care therapy is available, or who were not amenable to established forms of treatment.
2. Solid tumors must have measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
3. Female or male at 20 years of age or older.
4. ECOG performance status 0 to 2.
5. Recovered from prior treatment-related toxicity to at least grade 1 with exception of grade 2 alopecia.
6. Adequate organ function as defined by the following criteria:

   * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤3 x upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin ≤1.5 x ULN (except for subjects with documented Gilbert's syndrome)
   * Absolute neutrophil count (ANC) ≥ 1500/µL
   * Platelets ≥ 90,000/µL
   * Hemoglobin ≥ 9.0 g/dL
   * Serum creatinine ≤ 2.0 x ULN
7. Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

1. Major surgery or radiation therapy within 28 days of starting study treatment.
2. Systemic anti-cancer therapy within 28 days or 5 half-lives (whichever is shorter) of starting study treatment.
3. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
4. Current treatment on another clinical trial.
5. Spinal cord compression, carcinomatous meningitis, or leptomeningeal disease unless appropriately treated and neurologically stable for at least 4 weeks.
6. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack; within 6 months prior to starting study treatment for pulmonary embolus. However, upon agreement between the investigator and medical monitor, the 6-month post-event-free period for a subject with a pulmonary embolus can be waived if due to advanced cancer. Appropriate treatment with anticoagulants is permitted.
7. NYHA Class III or IV heart failure and known history of QTc prolongation or Torsade de Pointes.
8. Use of medications known to significantly prolong the QTc interval (e.g., anti-arrhythmic and psychotropic medications).
9. Hypertension that cannot be controlled by medications.
10. Current treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
11. Known human immunodeficiency virus (HIV)-positive and is receiving anti-retroviral therapy.
12. Positive test for hepatitis B (HBsAg) or hepatitis C (anti-HCV antibody).
13. History of receiving organ transplantation or immune disorders that require continuous immunosuppressant agent therapy.
14. Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to the use of effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
15. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that would impart, in the judgment of the investigator and/or medical monitor, excess risk associated with study participation or study drug administration, which would make the subject inappropriate for entry into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of NBM-BMX [Safety and Tolerability] | up to 28 days
  Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0
Maximum tolerated dose (MTD) of NBM-BMX [Safety and Tolerability] | up to 28 days
  The MTD will be defined as the dose level at which at most one of six patients experiences a DLT after 28 days of treatment have occurred, with the next higher dose having at least 2/3 or 2/6 patients experiencing a DLT.

SECONDARY OUTCOMES:
Preliminary assessment of anti-tumor activity by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) [Efficacy] | at least 8 weeks
AUC(0-last) of NBM-BMX [Pharmacokinetics] | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  AUC(0-last): area under the plasma concentration versus time curve to the time of the last measurable concentration
Cmax of NBM-BMX [Pharmacokinetics] | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  Cmax: maximum plasma concentration
Tmax of NBM-BMX [Pharmacokinetics] | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  Tmax: time to maximum plasma concentration
T(1/2) of NBM-BMX [Pharmacokinetics] | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  T(1/2): terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei